CLINICAL TRIAL: NCT02820012
Title: Multicenter Study on the Contribution of Surgical Treatment by ST2R Technique (Simultaneous Translation on Two Rods) in Scoliosis of the Children and Adolescents
Brief Title: Scoliosis Surgery - ST2R (Simultaneous Translation on Two Rods)
Acronym: ST2R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-HPNCL-01
Record Dates: First submitted 2016-05-31; First posted 2016-06-30 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Scoliosis
Keywords: Scoliosis; ST2R
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scoliosis (Other): Preoperative data: demographics, clinical diagnosis and etiology, relevant prior medical treatment, x-rays, and patient questionnaire will be completed in the database.
  The self-questionnaire (SAQ parents, patients, SR22) provided will assess the state of health and disability of patients.
  After surgery: the clinical questionnaire will be completed by the investigator to collect the parameters of the operation and the patient's clinical data Immediate Postoperative visit: J1 to S1: radiological and clinical examinations .
  Visit Month 1 to M3, M 12, M 24 , M 36 , M 60 : During these visits, clinical and radiological examinations will be realized.
  Interventions: Other: Scoliosis

INTERVENTIONS:
Other: Scoliosis — Questionnaires, radiography

SUMMARY:
Although practiced for many years, surgical correction of scoliosis is relatively subject published for idiopathic scoliosis and a few published for other types of scoliosis.

This study involves a creation of an observatory of patients undergoing scoliosis by ST2R reduction technique (Simultaneous Translation on Two Rods) associated with the PASS ® system.

The main objective is to analyze the three-dimensional correction of the deformity after intervention and its maintenance over time depending on the etiology of scoliosis.

This research is conducted in pediatric surgery services specialized in this technique.

Correcting radiographic parameters is directly related to the surgical procedure. The quality of life of patients is indirectly affected by the surgery. Secondary objectives are to analyze the surgical technique and to evaluate its impact on the quality of life of patients.

This study will firstly to have a better understanding in:

* Scoliosis of the children and adolescents and their surgical treatment;
* The impact of the surgical procedure by the ST2R technique on the three-dimensional correction, and the patient's quality of life; and secondly, better management of patients requiring surgery for scoliosis as well as a public health impact.

DETAILED DESCRIPTION:
The correction of the deformity in three planes of space is the main goal of surgical treatment of children's scoliosis and adolescents.

The techniques provide a satisfactory correction of the deformity in the coronal plane but remain insufficient in the sagittal plane and in particular for the correction of thoracic hypokyphosis.

Dr. Clarke and his team have shown that ST2R reduction technique (Simultaneous Translation on Two Rods) associated with the PASS ® system gave a good correction of the thoracic hypokyphosis of idiopathic scoliosis. The results of his single-center studies have shown that ST2R technique allowed to restore normal thoracic kyphosis with an average gain of 23 ° in patients preoperatively hypokyphosis, higher than the gains made by other techniques (rotation of the shaft, close off Gradually, in situ bending), while providing a frontal correction 70%, similar to results reported by other techniques. The results of this technique for non idiopathic scoliosis are still to be analyzed.

The creation of an observatory of children's and adolescents scoliosis (idiopathic, neuromuscular, etc ...) operated by the technique of reduction by simultaneous translation on two rods with the same instrumentation will:

* Firstly, to confirm or refute the first published results idiopathic scoliosis
* And secondly to analyze the results of the same technique on all other scoliosis.

The impact of the intervention on the quality of life of patients is an essential element that will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Scoliosis of the children and adolescents requiring surgical treatment by the technical ST2R
* Non-opposition form signed by the patient in a state to consent
* Non-opposition form signed by at least one of the legal representatives
* Children affiliated to the Social Security system

Exclusion Criteria:

* All cases that do not require surgical treatment by the technical ST2R
* Malformation or vertebral fractures
* All patients not willing to comply with instructions postoperative
* Opposition by the patient or legal guardian with the use of pre- and postoperative data
* Not affiliated to the Social Security system

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 164 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment radiographically of the dimensional scoliosis correction in the coronal plan | 60 months after chirurgical intervention
  Cobb angle measurements of curvatures

SECONDARY OUTCOMES:
Assessment of scoliosis in preoperative | baseline
  Cobb angles measurements of curvatures
Assessment radiographically of the dimensional scoliosis correction in the coronal plan | 5 minutes after the end of the chirurgical intervention
  Cobb angle measurements of curvatures
Assessment radiographically of the dimensional scoliosis correction in the sagittal plan | 5 minutes after the end of the chirurgical intervention
  angle of thoracic kyphosis vertebrae between T4 and T12
Assessment radiographically of the dimensional scoliosis correction in the axial plan | 5 minutes after the end of the chirurgical intervention
  measure of the vertebral rotation of the apical vertebra of the main curvature
Assessment of the postoperative complications | 60 month after the chirurgical intervention
  number of each postoperative complication
Assessment of the intra operative complications | 5 minutes after the end of the chirurgical intervention
  number of each intra operative complication
Assessment of the patient's quality of life | 60 month after the chirurgical intervention
  result to a self-administered questionnaire (SRS22)
Assessment radiographically of the dimensional scoliosis correction in the sagittal plan | 60 months after chirurgical intervention
  angle of thoracic kyphosis vertebrae between T4 and T12
Assessment radiographically of the dimensional scoliosis correction in the axial plan | 60 months after chirurgical intervention
  measure of the vertebral rotation of the apical vertebra of the main curvature

CONTACTS AND LOCATIONS:
Overall Officials: Frederico Solla, MD, Principal Investigator — Fondation Lenval
Locations (5):
- France (5):
  - Hôpital Jean Minjoz, CHU Besançon, Besançon
  - Hôpital Femme Mère Enfant, Bron
  - Centre Orthopédique Santy, Lyon
  - Hôpital mère-enfant pédiatrie, CHU Nantes, Nantes
  - Hôpitaux Pédiatriques CHU-LENVAL, Nice

IPD SHARING:
Plan to Share IPD: No